CLINICAL TRIAL: NCT04692012
Title: Successful Treatment of Residual Hypermetropic Refraction on Pseudophakic Patients Using Allogenic Fresh Myopic Lenticule Implantation with ReLex-Smile Surgery
Brief Title: Treatment of Residual Hypermetropic Refraction on Pseudophakic Patients Using Allogenic Fresh Myopic Lenticule
Acronym: ReLex-Smile
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHPristina
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pseudophakia; Hypermetropia; Myopia
MeSH Terms: conditions — Pseudophakia; Hyperopia; Myopia

STUDY DESIGN:
Intervention Model Description: pseudophakic group hyperopic group myopic group
Masking Description: pseudophakic (Trifocal IOL) group 492 patients-246 eyes residual hyperopic group 34 patients-38 eyes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FRESH CORNEAL LENTICULE IMPLANTATION (Other): The aim of this study is to investigate the effect of fresh corneal myopic lenticule implantation as allogenic implant that will be taken from myopic patients to implant on pseudophakic patients with residual hypermetropic refraction using VisuMax Femtosecond Laser-Smile module surgery with primary objective to assess(increase) visual acuity.
  Interventions: Other: FRESH CORNEAL MYOPIC LENTICULE IMPLANTATION

INTERVENTIONS:
Other: FRESH CORNEAL MYOPIC LENTICULE IMPLANTATION — VisuMax femtosecond laser performed flap-cut procedure with an energy cut index of 30 nJ (150nJ), spot and track spacing surface cut of 4.5 μm, side cut 2.0 μm were used to create an intrastromal pocket into the patient's cornea to receive the donor lenticule. The stromal pocket diameter was set 7.6 to 8.0 mm (1 mm larger than the optical zone of the donor lenticule) and cap thickness was set to 130 μm from corneal surface and a 4 mm superior incision. Hinge position flap was set at 90°, angle 50° and width 4 mm, side cut angle 90°. The pocket was dissected using a blunt spatula washed with normal saline. The lenticule was held with lenticule forceps and gently inserted into the pocket through the 4 mm superior incision. Incision position changed according to the position of the highest K values. Current orientation was marked with a sterile skin marker. The lenticule was positioned around the marked center of the cone and flattened out from the surface using a blunt spatula.
  Other Names: Relex smile surgery

SUMMARY:
The residual hypermetropic refraction on pseudophakic(Trifocal IOL) patients is difficult to treat surgically. In addition, there are not many suitable options to offer such patients presenting with this condition.

Two current common surgeries to treat residual hyperopic refraction are refractive lens exchange (RLE) and excimer laser ablation (LASIK or PRK).

Laser procedures: Photorefractive keratectomy (PRK); Laser assisted in situ keratomileusis (LASIK); Risks of LASIK include abnormalities of the corneal flap, epithelial ingrowth, corneal ectasia, refractive surprises, irregular astigmatism, decentration, visual aberrations, a loss of BCVA, infectious keratitis, symptoms, and diffuse lamellar keratitis.

Refractive lens exchange (RLE); The risks of RLE are similar to those of cataract surgery and include endophthalmitis, a loss of accommodation, vitreous loss with posterior capsular rupture, and retinal detachment.

The method used at the EYE Hospital Pristina using fresh lenticule implantation by ReLex-SMILE is safe and effective method, since there is no flap this prevents invasive damage to the anterior surface of the cornea contrary to the LASIK where flap is present posing risk for epithelial ingrowth.

Before SMILE,YAG-laser capsulotomy should be performed on all patients, regardless of posterior capsule ossification, in pseudophakic patients with residual refraction. When the YAG-laser is applied after the SMILE,there will be a diopter change.

DETAILED DESCRIPTION:
This study is to investigate the effect of fresh myopic corneal lenticule implantation as allogenic implant that will be taken from myopic patients to implant on pseudophakic patients(Trifocal IOL) with residual hypermetropic refraction(over +0.50Dsph) using VisuMax Femtosecond laser - Smile module surgery with primary objective to assess (increase) visual acuity . In pseudophakic patients with hyperopic astigmatism residual refraction, corneal topography-guided intrastromal fresh lenticule implantation should be performed and the lenticule was placed according to the low K value.

ELIGIBILITY:
Inclusion Criteria:

* residual hypermetropic refraction on pseudophakic patients
* low visual acuity

Exclusion Criteria:

* active anterior segment pathologic features,
* previous corneal or anterior segment surgery,
* glaucoma,
* retinal detachment

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
increasing of visual acuity | 12 months
  using fresh myopic corneal lenticule for treatment of residual hypermetropic refraction on pseudophakic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo